CLINICAL TRIAL: NCT03926169
Title: A Phase 2, Multicenter, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Safety and Efficacy of Risankizumab in Adult Subjects With Moderate to Severe Hidradenitis Suppurativa
Brief Title: A Global Study Comparing Risankizumab to Placebo in Adult Participants With Moderate to Severe Hidradenitis Suppurativa
Acronym: DETERMINED 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M16-833; 2019-000122-21 (EudraCT Number)
Record Dates: First submitted 2019-04-23; First posted 2019-04-24 (Actual); Results first posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-07

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa; Risankizumab; Placebo
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Risankizumab 180 mg (Experimental): In Period A, participants receive blinded risankizumab 180 mg via a subcutaneous (SC) injection at Weeks 0 (Baseline), 1, 2, 4, and 12.
  Interventions: Drug: Risankizumab
- Risankizumab 360 mg (Experimental): In Period A, participants receive blinded risankizumab 360 mg via a SC injection at Weeks 0 (Baseline), 1, 2, 4, and 12.
  Interventions: Drug: Risankizumab
- Placebo (Placebo Comparator): In Period A, participants receive blinded placebo via a SC injection at Weeks 0 (Baseline), 1, 2, 4, and 12.
  Interventions: Drug: Placebo for risankizumab
- Risankizumab 180 mg / Risankizumab 360 mg (Experimental): In Period A, participants receive blinded risankizumab 180 mg via a subcutaneous (SC) injection at Weeks 0 (Baseline), 1, 2, 4, and 12.
  In Period B, participants receive blinded placebo at Weeks 16, 17, and 18. Starting at Week 20, participants receive open-label risankizumab 360 mg every 8 weeks (q8w) at Weeks 20, 28, 36, 44, 52, and 60.
  Interventions: Drug: Risankizumab; Drug: Placebo for risankizumab
- Risankizumab 360 mg / Risankizumab 360 mg (Experimental): In Period A, participants receive blinded risankizumab 360 mg via a SC injection at Weeks 0 (Baseline), 1, 2, 4, and 12.
  In Period B, participants receive blinded placebo at Weeks 16, 17, and 18. Starting at Week 20, participants receive open-label risankizumab 360 mg q8w at Weeks 20, 28, 36, 44, 52, and 60.
  Interventions: Drug: Risankizumab; Drug: Placebo for risankizumab
- Placebo / Risankizumab 360 mg (Placebo Comparator): In Period A, participants receive blinded placebo via a SC injection at Weeks 0 (Baseline), 1, 2, 4, and 12.
  In Period B, participants receive blinded risankizumab 360 mg at Weeks 16, 17, and 18. Starting at Week 20, participants receive open-label risankizumab 360 mg q8w at Weeks 20, 28, 36, 44, 52, and 60.
  Interventions: Drug: Risankizumab; Drug: Placebo for risankizumab

INTERVENTIONS:
Drug: Risankizumab — Risankizumab is administered as a SC injection in pre-filled syringe (PFS)
  Other Names: ABBV-066; SKYRIZI
  Arms: Placebo / Risankizumab 360 mg; Risankizumab 180 mg; Risankizumab 180 mg / Risankizumab 360 mg; Risankizumab 360 mg; Risankizumab 360 mg / Risankizumab 360 mg
Drug: Placebo for risankizumab — Placebo for risankizumab is administered as a SC injection in PFS
  Arms: Placebo; Placebo / Risankizumab 360 mg; Risankizumab 180 mg / Risankizumab 360 mg; Risankizumab 360 mg / Risankizumab 360 mg

SUMMARY:
The primary objective of this study is to assess the safety and efficacy of risankizumab 180 mg and 360 mg versus placebo for the treatment of signs and symptoms of moderate to severe hidradenitis suppurativa (HS) in adult participants diagnosed for at least one year before the Baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Participant with moderate to severe HS for at least 1 year prior to baseline visit.
* HS lesions present in at least two distinct anatomical areas.
* Draining fistula count of ≤ 20 at Baseline visit.
* Total abscess and inflammatory nodule (AN) count of ≥ 5 at Baseline visit.
* Participants are required to use a daily antiseptic wash on their HS lesions.
* Participant must have a history of inadequate response or intolerance to an adequate trial of oral antibiotics for treatment of HS.

Exclusion Criteria:

* Participant has a history of active skin disease other than HS that could interfere with the assessment of HS.
* Participant has active tuberculosis (TB) or concurrent treatment for latent TB or evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV) or human immunodeficiency virus (HIV) infection.
* Participant has prior exposure to anti-interleukin-1 (anti-IL-1) treatment within 3 months or 5 half-lives, whichever is longer, prior to baseline.
* Participant has received prescription topical therapies (including topical antibiotics) within 14 days prior to the Baseline visit.
* Participant has received systemic non-biologic therapies that can also be used to treat HS within 4 weeks prior to the Baseline visit.
* Participant has received any systemic (including oral) antibiotic treatment within 4 weeks prior to the Baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (59):
- United States (22):
  - Burke Pharmaceutical Research /ID# 211671, Hot Springs, Arkansas
  - Bakersfield Derma & Skin Cance /ID# 211684, Bakersfield, California
  - Wallace Medical Group /ID# 215958, Los Angeles, California
  - Integrative Skin Science and Research /ID# 212550, Sacramento, California
  - UC Davis Health /ID# 211436, Sacramento, California
  - California Dermatology Institute /ID# 211786, Thousand Oaks, California
  - CCD Research, PLLC /ID# 214479, Cromwell, Connecticut
  - Advanced Medical Research /ID# 215203, Sandy Springs, Georgia
  - Arlington Dermatology /ID# 219096, Rolling Meadows, Illinois
  - Tufts Medical Center /ID# 212680, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center /ID# 211794, Boston, Massachusetts
  - Hamzavi Dermatology /ID# 212318, Fort Gratiot, Michigan
  - University of Minnesota /ID# 212319, Minneapolis, Minnesota
  - Minnesota Clinical Study Center /ID# 211979, New Brighton, Minnesota
  - Skin Specialists, PC /ID# 211675, Omaha, Nebraska
  - Montefiore Medical Center - Moses Campus /ID# 211800, The Bronx, New York
  - Oregon Medical Res Center PC /ID# 211796, Portland, Oregon
  - Penn State Hershey Medical Ctr /ID# 211659, Hershey, Pennsylvania
  - Rhode Island Hospital /ID# 211807, Providence, Rhode Island
  - Modern Research Associates, PL /ID# 215202, Dallas, Texas
  - Virginia Clinical Research, Inc. /ID# 215959, Norfolk, Virginia
  - Premier Clinical Research /ID# 211799, Spokane, Washington
- Australia (7):
  - Woden Dermatology /ID# 212437, Phillip, Australian Capital Territory
  - Westmead Hospital /ID# 212438, Westmead, New South Wales
  - Veracity Clinical Research /ID# 212432, Woolloongabba, Queensland
  - Skin Health Institute Inc /ID# 212433, Carlton, Victoria
  - Sinclair Dermatology /ID# 215548, East Melbourne, Victoria
  - The Royal Melbourne Hospital /ID# 212436, Parkville, Victoria
  - Fremantle Dermatology /ID# 212434, Fremantle, Western Australia
- Canada (5):
  - Wiseman Dermatology Research /ID# 212243, Winnipeg, Manitoba
  - Dr. Irina Turchin PC Inc. /ID# 212248, Fredericton, New Brunswick
  - Dr. S.K. Siddha Medicine Professional Corporation /ID# 219043, Newmarket, Ontario
  - K. Papp Clinical Research /ID# 212166, Waterloo, Ontario
  - Dre Angelique Gagne-Henley M.D. inc. /ID# 212249, Saint-Jérôme, Quebec
- France (6):
  - Chu de Nice-Hopital L'Archet Ii /Id# 212563, Nice, Alpes-Maritimes
  - CHU de SAINT ETIENNE - Hopital Nord /ID# 212564, Saint Priest EN Jarez, Pays de la Loire Region
  - HCL - Hopital Edouard Herriot /ID# 218408, Lyon
  - Polyclinique Courlancy /ID# 212567, Reims
  - CHU Toulouse - Hopital Larrey /ID# 213581, Toulouse
  - Hopital Prive d'Antony /ID# 212566, Antony, Île-de-France Region
- Germany (4):
  - Universitaetsklinikum Frankfurt /ID# 211913, Frankfurt am Main, Hesse
  - Klinikum Ruhr Univ Bochum /ID# 211910, Bochum
  - Staedtisches Klinikum Dessau /ID# 211914, Dessau
  - Universitaetsklinikum Hamburg-Eppendorf (UKE) /ID# 211912, Hamburg
- Japan (5):
  - Nagoya City University Hospital /ID# 211155, Nagoya, Aichi-ken
  - Fukuoka University Hospital /ID# 211303, Fukuoka, Fukuoka
  - Tohoku University Hospital /ID# 212214, Sendai, Miyagi
  - University of the Ryukyus Hospital /ID# 211373, Nakagami-gun, Okinawa
  - Toranomon Hospital /ID# 211742, Minato-ku, Tokyo
- Netherlands (3):
  - Bravis Ziekenhuis /ID# 212536, Bergen op Zoom, North Brabant
  - Erasmus Medisch Centrum /ID# 212535, Rotterdam, South Holland
  - Amphia Ziekenhuis /ID# 212538, Breda
- Spain (7):
  - Consorci Corporacio Sanitaria Parc Tauli Sabadell /ID# 212015, Sabadell, Barcelona
  - Hospital de Manises /ID# 211541, Manises, Valencia
  - Hospital General Universitario Alicante /ID# 212010, Alicante
  - Hospital Santa Creu i Sant Pau /ID# 212009, Barcelona
  - Hospital Universitario Virgen de las Nieves /ID# 212014, Granada
  - Hospital General Universitario Gregorio Maranon /ID# 212011, Madrid
  - Hospital Universitario Virgen de la Victoria /ID# 212013, Málaga

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Kimball AB, Prens EP, Passeron T, Maverakis E, Turchin I, Beeck S, Drogaris L, Geng Z, Zhan T, Messina I, Bechara FG. Efficacy and Safety of Risankizumab for the Treatment of Hidradenitis Suppurativa: A Phase 2, Randomized, Placebo-Controlled Trial. Dermatol Ther (Heidelb). 2023 May;13(5):1099-1111. doi: 10.1007/s13555-023-00913-3. Epub 2023 Mar 9. PMID 36892753
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In Period A, participants who met the study's eligibility criteria were randomized at the Baseline Visit, in a 1:1:1 ratio, to receive either placebo, risankizumab 180 mg or 360 mg via a subcutaneous (SC) injection.
Groups:
- Placebo / Risankizumab 360 mg: In Period A, participants received blinded placebo via SC injection at Weeks 0 (Baseline), 1, 2, 4, and 12.
  In Period B, participants received blinded risankizumab 360 mg at Weeks 16, 17, and 18. Starting at Week 20, participants received open-label risankizumab 360 mg every 8 weeks (q8w) at Weeks 20, 28, 36, 44, 52, and 60.
- Risankizumab 180 mg / Risankizumab 360 mg: In Period A, participants received blinded risankizumab 180 mg via SC injection at Weeks 0 (Baseline), 1, 2, 4, and 12.
  In Period B, participants received blinded placebo at Weeks 16, 17, and 18. Starting at Week 20, participants received open-label risankizumab 360 mg q8w at Weeks 20, 28, 36, 44, 52, and 60.
- Risankizumab 360 mg / Risankizumab 360 mg: In Period A, participants received blinded risankizumab 360 mg via SC injection at Weeks 0 (Baseline), 1, 2, 4, and 12.
  In Period B, participants received blinded placebo at Weeks 16, 17, and 18. Starting at Week 20, participants received open-label risankizumab 360 mg q8w at Weeks 20, 28, 36, 44, 52, and 60.
Period: Period A
Arm/Group | Placebo / Risankizumab 360 mg | Risankizumab 180 mg / Risankizumab 360 mg | Risankizumab 360 mg / Risankizumab 360 mg
Started (Randomized) | 82 | 80 | 81
Never Received Study Drug | 0 | 0 | 1
Completed (Completed Week 16) | 74 | 70 | 75
Not Completed | 8 | 10 | 6
Not completed — Adverse Event | 2 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 2
Not completed — Lost to Follow-up | 3 | 1 | 0
Not completed — Lack of Efficacy | 0 | 2 | 2
Not completed — COVID-19 Infection | 0 | 1 | 0
Not completed — COVID-19 Logistical Restrictions | 0 | 2 | 1
Not completed — Other, Not Specified | 1 | 0 | 0
Period: Period B
Arm/Group | Placebo / Risankizumab 360 mg | Risankizumab 180 mg / Risankizumab 360 mg | Risankizumab 360 mg / Risankizumab 360 mg
Started (Entered Period B) | 74 | 70 | 75
Entered Period B and Received Study Drug | 74 | 70 | 74
Completed (Completed study) | 4 | 7 | 4
Not Completed | 70 | 63 | 71
Not completed — Adverse Event | 3 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 3 | 0
Not completed — Lack of Efficacy | 3 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 4
Not completed — Other, Not Specified | 62 | 57 | 65

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo / Risankizumab 360 mg | Risankizumab 180 mg / Risankizumab 360 mg | Risankizumab 360 mg / Risankizumab 360 mg | Total
Number analyzed (Participants) | 82 | 80 | 81 | 243
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (11.97) | 38.9 (11.45) | 38.2 (11.99) | 38.1 (11.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 53 | 51 | 152
  Male | 34 | 27 | 30 | 91
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 7 | 26
  Not Hispanic or Latino | 73 | 70 | 74 | 217
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 68 | 63 | 62 | 193
  Black or African American | 4 | 12 | 9 | 25
  Asian | 8 | 4 | 9 | 21
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Multiple Races | 2 | 0 | 1 | 3
Abscess and Inflammatory Nodule (AN) Count [Mean (Standard Deviation); unit: abscess and inflammatory nodules] | 15.7 (28.42) | 13.7 (11.42) | 12.5 (8.24) | 14.0 (18.36)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Hidradenitis Suppurativa Clinical Response (HiSCR) at Week 16
Description: HiSCR is defined as at least a 50% reduction from Baseline in the total abscess and inflammatory nodule (AN) count, with no increase in abscess or draining fistula counts.
Time Frame: Baseline (Week 0), Week 16
Population: Intent-to-Treat Population: all randomized participants. Non-responder imputation with multiple imputation to handle missing data due to COVID-19 (NRI-C) .
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Groups:
- Placebo: In Period A, participants received blinded placebo via SC injection at Weeks 0 (Baseline), 1, 2, 4, and 12.
- Risankizumab 180 mg: In Period A, participants received blinded risankizumab 180 mg via SC injection at Weeks 0 (Baseline), 1, 2, 4, and 12.
- Risankizumab 360 mg: In Period A, participants received blinded risankizumab 360 mg via SC injection at Weeks 0 (Baseline), 1, 2, 4, and 12.
Arm/Group | Placebo | Risankizumab 180 mg | Risankizumab 360 mg
Number analyzed (Participants) | 82 | 80 | 81
percentage of participants | 41.5 [29.3 to 53.7] | 46.8 [34.2 to 59.4] | 43.4 [31.0 to 55.8]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 180 mg; Test type: Superiority; p = 0.422, Cochran-Mantel-Haenszel — Across the strata, 97.5% confidence interval for adjusted difference and P-value were calculated according to the Cochran-Mantel-Haenszel test adjusted for the actual values stratification factors under a two-sided alpha level 0.025 for each dose; Adjusted Response Rate Difference (%) = 6.0, 97.5% CI 2-sided [-10.8 to 22.8]
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 360 mg; Test type: Superiority; p = 0.858, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted Response Rate Difference (%) = 1.3, 97.5% CI 2-sided [-15.4 to 18.1]

2. Secondary Outcome: Percentage of Participants Achieving ≥ 30% Reduction and ≥ 1 Unit Reduction From Baseline in Patient's Global Assessment (PGA) of Skin Pain Numerical Rating Scale (NRS30) at Week 8 Among Participants With Baseline Numerical Rating Scale (NRS) ≥ 3
Description: NRS30 is evaluated based on worst skin pain in a 24-hour recall period (maximal daily pain), ranging from 0 (no skin pain) to 10 (skin pain as bad as you can imagine). The percentage of participants who achieved at least 30% reduction and at least 1 unit reduction from Baseline at Week 8 in the PGA of Skin Pain (NRS30) - at worst, among participants with Baseline NRS ≥ 3, is presented.
Time Frame: Baseline (Week 0) to Week 8
Population: Intent-to-Treat Population: all randomized participants. Participants with Baseline NRS ≥ 3. Non-responder imputation with multiple imputation to handle missing data due to COVID-19.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab 180 mg | Risankizumab 360 mg
Number analyzed (Participants) | 61 | 61 | 60
percentage of participants | 33.0 [19.4 to 46.5] | 29.2 [15.9 to 42.6] | 40.0 [25.8 to 54.2]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 180 mg; Test type: Superiority; p = 0.725, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted Response Rate Difference (%) = -3.0, 97.5% CI 2-sided [-21.8 to 15.9]
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 360 mg; Test type: Superiority; p = 0.301, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted Response Rate Difference (%) = 8.8, 97.5% CI 2-sided [-10.3 to 27.8]

3. Secondary Outcome: Percentage of Participants Achieving ≥ 30% Reduction and ≥ 1 Unit Reduction From Baseline in PGA of Skin Pain Numerical Rating Scale (NRS30) at Week 16 Among Participants With Baseline Numerical Rating Scale (NRS) ≥ 3
Description: NRS30 is evaluated based on worst skin pain in a 24-hour recall period (maximal daily pain), ranging from 0 (no skin pain) to 10 (skin pain as bad as you can imagine). The percentage of participants who achieved at least 30% reduction and at least 1 unit reduction from Baseline at Week 16 in the PGA of Skin Pain (NRS30) - at worst, among participants with Baseline NRS ≥ 3, is presented.
Time Frame: Baseline (Week 0) to Week 16
Population: as for outcome 2
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab 180 mg | Risankizumab 360 mg
Number analyzed (Participants) | 61 | 61 | 60
percentage of participants | 27.9 [15.0 to 40.7] | 31.1 [17.5 to 44.7] | 38.6 [24.4 to 52.7]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 180 mg; Test type: Superiority; p = 0.650, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted Response Rate Difference (%) = 3.7, 97.5% CI 2-sided [-14.5 to 21.8]
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 360 mg; Test type: Superiority; p = 0.147, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted Response Rate Difference (%) = 12.3, 97.5% CI 2-sided [-6.7 to 31.3]

4. Secondary Outcome: Percentage of Participants Who Experienced ≥ 25% Increase in Abscess and Inflammatory Nodule (AN) Counts in Period A With a Minimum Increase of 2 Relative to Baseline
Time Frame: Baseline (Week 0) to Week 16
Population: Intent-to-Treat Population: all randomized participants. Participants with Baseline NRS ≥ 3. Non-responder imputation.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Risankizumab 180 mg | Risankizumab 360 mg
Number analyzed (Participants) | 82 | 80 | 81
percentage of participants | 29.3 [18.0 to 40.5] | 22.5 [12.0 to 33.0] | 18.5 [8.8 to 28.2]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 180 mg; Test type: Superiority; p = 0.342, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted Response Rate Difference (%) = -6.5, 97.5% CI 2-sided [-21.8 to 8.8]
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 360 mg; Test type: Superiority; p = 0.108, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted Response Rate Difference (%) = -10.6, 97.5% CI 2-sided [-25.3 to 4.2]

5. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Week 16
Description: The DLQI is a 10-item validated questionnaire used to assess the impact of HS disease symptoms and treatment on quality of life (QoL). It consists of 10 questions evaluating impact of skin diseases on different aspects of a participant's QoL over the prior week, including symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the side effects of treatment. DLQI scores range from 0 to 30, with a higher score indicating a more impaired QoL.
Time Frame: Baseline (Week 0) to Week 16
Population: Intent-to-Treat Population: all randomized participants. Participants with an assessment at given time point.
Measure: Least Squares Mean (97.5% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Risankizumab 180 mg | Risankizumab 360 mg
Number analyzed (Participants) | 62 | 66 | 63
score on a scale | -2.1 [-3.9 to -0.4] | -3.5 [-5.2 to -1.8] | -3.7 [-5.5 to -2.0]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 180 mg; Test type: Superiority; p = 0.179, mixed-effect model repeat measures — Mixed-effect model repeat measures analysis with treatment, visit, treatment by visit interaction, stratification factor and baseline measurement in the model. An unstructured variance covariance matrix is used; LS Mean Difference = -1.3, 97.5% CI 2-sided [-3.5 to 0.9], Standard Error of Mean 0.97
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 360 mg; Test type: Superiority; p = 0.105, mixed-effect model repeat measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -1.6, 97.5% CI 2-sided [-3.8 to 0.6], Standard Error of Mean 0.98

6. Secondary Outcome: Change From Baseline in HS-Related Swelling Based on the Hidradenitis Suppurativa Symptom Assessment (HSSA) Swollen Skin Score at Week 16
Description: HSSA is a 9-item participant-reported outcome (PRO) questionnaire developed to assess the symptoms of HS. HS-related swelling is scored on an 11-point NRS, where 0 represents no symptoms and 10 represents extreme symptom experience.
Time Frame: Baseline (Week 0) to Week 16
Population: Intent-to-Treat Population: all randomized participants. Participants with an assessment at given time point.
Measure: Least Squares Mean (97.5% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Risankizumab 180 mg | Risankizumab 360 mg
Number analyzed (Participants) | 65 | 53 | 63
score on a scale | -0.870 [-1.416 to -0.324] | -0.751 [-1.338 to -0.165] | -0.885 [-1.436 to -0.334]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 180 mg; Test type: Superiority; p = 0.727, mixed-effect model repeat measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = 0.118, 97.5% CI 2-sided [-0.646 to 0.883], Standard Error of Mean 0.3385
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 360 mg; Test type: Superiority; p = 0.963, mixed-effect model repeat measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -0.015, 97.5% CI 2-sided [-0.755 to 0.724], Standard Error of Mean 0.3273

7. Secondary Outcome: Change From Baseline in HS-Related Odor Based on the HSSA Bad Smell Score at Week 16
Description: HSSA is a 9-item PRO questionnaire developed to assess the symptoms of HS. HS-related odor is scored on an 11-point NRS, where 0 represents no symptoms and 10 represents extreme symptom experience.
Time Frame: Baseline (Week 0) to Week 16
Population: Intent-to-Treat Population: all randomized participants. Participants with an assessment at given time point.
Measure: Least Squares Mean (97.5% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Risankizumab 180 mg | Risankizumab 360 mg
Number analyzed (Participants) | 65 | 53 | 63
score on a scale | -0.677 [-1.160 to -0.195] | -0.635 [-1.149 to -0.120] | -0.442 [-0.928 to 0.044]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 180 mg; Test type: Superiority; p = 0.886, mixed-effect model repeat measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = 0.042, 97.5% CI 2-sided [-0.622 to 0.706], Standard Error of Mean 0.2941
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 360 mg; Test type: Superiority; p = 0.409, mixed-effect model repeat measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = 0.236, 97.5% CI 2-sided [-0.408 to 0.879], Standard Error of Mean 0.2851

8. Secondary Outcome: Change From Baseline in HS-Related Worst Drainage Based on the HSSA Worst Drainage Score at Week 16
Description: HSSA is a 9-item PRO questionnaire developed to assess the symptoms of HS. HS-related worst drainage is scored on an 11-point NRS, where 0 represents no symptoms and 10 represents extreme symptom experience.
Time Frame: Baseline (Week 0) to Week 16
Population: Intent-to-Treat Population: all randomized participants. Participants with an assessment at given time point.
Measure: Least Squares Mean (97.5% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Risankizumab 180 mg | Risankizumab 360 mg
Number analyzed (Participants) | 65 | 53 | 63
score on a scale | -0.630 [-1.154 to -0.107] | -0.882 [-1.440 to -0.324] | -0.705 [-1.233 to -0.176]
Statistical Analysis 1: Comparison: Placebo vs Risankizumab 180 mg; Test type: Superiority; p = 0.434, mixed-effect model repeat measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -0.252, 97.5% CI 2-sided [-0.977 to 0.473], Standard Error of Mean 0.3212
Statistical Analysis 2: Comparison: Placebo vs Risankizumab 360 mg; Test type: Superiority; p = 0.813, mixed-effect model repeat measures — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -0.074, 97.5% CI 2-sided [-0.779 to 0.631], Standard Error of Mean 0.3123

ADVERSE EVENTS:
Time Frame: From the first dose of study medication until 20 weeks after the last dose. Part A overall mean duration on study drug was 108.5 days. Part B overall mean duration on study drug was 179.9 days.
Groups:
- Placebo: In Period A, participants received blinded placebo via a SC injection at Weeks 0 (Baseline), 1, 2, 4, and 12.
- Risankizumab 180 mg: In Period A, participants received blinded risankizumab 180 mg via a SC injection at Weeks 0 (Baseline), 1, 2, 4, and 12.
- Risankizumab 360 mg: In Period A, participants received blinded risankizumab 360 mg via a SC injection at Weeks 0 (Baseline), 1, 2, 4, and 12.
- Placebo / Risankizumab 360 mg: In Period A, participants received blinded placebo via a SC injection at Weeks 0 (Baseline), 1, 2, 4, and 12.
  In Period B, participants received blinded risankizumab 360 mg at Weeks 16, 17, and 18. Starting at Week 20, participants received open-label risankizumab 360 mg every 8 weeks (q8w) at Weeks 20, 28, 36, 44, 52, and 60.
- Risankizumab 180 mg / Risankizumab 360 mg: In Period A, participants received blinded risankizumab 180 mg via a SC injection at Weeks 0 (Baseline), 1, 2, 4, and 12.
  In Period B, participants received blinded placebo at Weeks 16, 17, and 18. Starting at Week 20, participants received open-label risankizumab 360 mg q8w at Weeks 20, 28, 36, 44, 52, and 60.
- Risankizumab 360 mg / Risankizumab 360 mg: In Period A, participants received blinded risankizumab 360 mg via a SC injection at Weeks 0 (Baseline), 1, 2, 4, and 12.
  In Period B, participants received blinded placebo at Weeks 16, 17, and 18. Starting at Week 20, participants received open-label risankizumab 360 mg q8w at Weeks 20, 28, 36, 44, 52, and 60.
Arm/Group | Placebo | Risankizumab 180 mg | Risankizumab 360 mg | Placebo / Risankizumab 360 mg | Risankizumab 180 mg / Risankizumab 360 mg | Risankizumab 360 mg / Risankizumab 360 mg
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/80 | 0/80 | 0/74 | 0/70 | 0/74
Serious Adverse Events (participants affected / at risk) | 2/82 | 3/80 | 2/80 | 3/74 | 4/70 | 0/74
Other Adverse Events (participants affected / at risk) | 19/82 | 21/80 | 26/80 | 26/74 | 12/70 | 19/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=82) | Risankizumab 180 mg (N=80) | Risankizumab 360 mg (N=80) | Placebo / Risankizumab 360 mg (N=74) | Risankizumab 180 mg / Risankizumab 360 mg (N=70) | Risankizumab 360 mg / Risankizumab 360 mg (N=74)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TONSILLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
AFFECTIVE DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INTENTIONAL SELF-INJURY (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MAJOR DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ENDOMETRIOSIS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OVARIAN CYST (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HIDRADENITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABORTION INDUCED (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=82) | Risankizumab 180 mg (N=80) | Risankizumab 360 mg (N=80) | Placebo / Risankizumab 360 mg (N=74) | Risankizumab 180 mg / Risankizumab 360 mg (N=70) | Risankizumab 360 mg / Risankizumab 360 mg (N=74)
DIARRHOEA (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (4) | 5 (5) | 1 (1) | 2 (2)
NASOPHARYNGITIS (Infections and infestations) | 3 (3) | 6 (6) | 7 (8) | 1 (1) | 4 (5) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 4 (4) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 4 (4) | 2 (2) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 9 (16) | 6 (6) | 11 (15) | 7 (10) | 1 (1) | 4 (5)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 4 (4)
HIDRADENITIS (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (3) | 2 (3) | 6 (6) | 8 (8) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/69/NCT03926169/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT03926169/SAP_001.pdf